CLINICAL TRIAL: NCT00004859
Title: A Randomized Phase III Trial of Carboplatin, Paclitaxel and Thoracic Radiotherapy, With or Without Thalidomide, in Patients With Stage III Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Carboplatin, Paclitaxel, and Radiation Therapy With or Without Thalidomide in Patients With Stage III Non-small Cell Lung Cancer
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Trial was stopped early for futility
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02943; U10CA021115 (NIH); E3598 (Other: Eastern Cooperative Oncology Group (ECOG)); CDR0000067510 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2000-03-07; First posted 2003-01-27 (Estimated); Results first posted 2012-03-22 (Estimated); Last update posted 2014-06-02 (Estimated); Status verified 2013-02

CONDITIONS: Lung Cancer
Keywords: squamous cell lung cancer; large cell lung cancer; stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer; adenocarcinoma of the lung; adenosquamous cell lung cancer; bronchoalveolar cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Adenocarcinoma of Lung; Adenocarcinoma, Bronchiolo-Alveolar | interventions — Carboplatin; Paclitaxel; Thalidomide; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A (Paclitaxel + Carboplatin + RT) (Active Comparator): Induction chemotherapy dosing: Paclitaxel, 225 mg/m² (3 hour infusion) Day 1. Carboplatin, area under the plasma drug concentration versus time curve (AUC) =6.0, 15-30 min IV infusion immediately following paclitaxel, Day 1
  Concurrent chemotherapy / radiotherapy dosing: Paclitaxel, 45 mg/m2, administered weekly during radiotherapy over one hour. Carboplatin, AUC=2, 15- 30 minutes IV infusion immediately following paclitaxel; administered weekly during radiotherapy
  Radiation therapy started between days 43-50 from day 1 of cycle 1. The primary tumor and areas of known nodal disease received 60 Gy at 2.0 Gy fractions, 5 fractions/week for 30 fractions over 6 weeks to the post chemotherapy tumor volume as seen on computed tomography (CT). The initial 50 Gy was delivered to target volume (TV). The final 10 Gy was delivered to a reduced volume targeting defined by TV
  Interventions: Drug: carboplatin; Drug: paclitaxel; Radiation: radiation therapy
- Arm B (Paclitaxel + Carboplatin + RT+ Thalidomide) (Experimental): paclitaxel, carboplatin, and radiotherapy are same as those in Arm A.
  thalidomide: Induction chemotherapy dosing, oral daily, starting Day 1 for 24 months or until disease progression. Concurrent chemotherapy / radiotherapy dosing, oral daily, begin with 200 mg thalidomide as a single dose at bedtime. The dose is then increased by 100 mg every week as tolerated up to a total dose of 1000 mg.
  Interventions: Drug: carboplatin; Drug: paclitaxel; Drug: thalidomide; Radiation: radiation therapy

INTERVENTIONS:
Drug: carboplatin — Induction Chemotherapy dosing: AUC=6.0, 15-30 min IV infusion immediately following paclitaxel, Day 1 and Day 22. Concurrent Chemotherapy / Radiotherapy dosing, AUC=2; 15- 30 minutes IV infusion immediately following paclitaxel; administered weekly during radiotherapy
  Other Names: CBDCA; Paraplatin; JM-8; NSC 241240
Drug: paclitaxel — Induction chemotherapy dosing: 225 mg/m² (3 hour infusion) Day 1 and Day 22. Concurrent Chemotherapy / Radiotherapy dosing: 45 mg/m2; administered weekly during radiotherapy over one hour
  Other Names: Taxol; NSC 125973
Drug: thalidomide — Induction Chemotherapy dosing: oral daily, starting Day 1 for 24 months or until disease progression. Concurrent Chemotherapy / Radiotherapy dosing: oral daily, begin with 200 mg thalidomide as a single dose at bedtime. The dose is then increased by 100 mg every week as tolerated up to a total dose of 1000 mg.
  Other Names: (d,1)-N phthalidoglutarimide; Thalomid; NSC #66847; IND # 48832
  Arms: Arm B (Paclitaxel + Carboplatin + RT+ Thalidomide)
Radiation: radiation therapy — Radiation therapy started between days 43-50 from day 1 of cycle 1. The primary tumor and areas of known nodal disease received 60 Gy at 2.0 Gy fractions, 5 fractions/week for 30 fractions over 6 weeks to the post chemotherapy tumor volume as seen on computed tomography (CT). The initial 50 Gy was delivered to target volume (TV). The final 10 Gy was delivered to a reduced volume targeting defined by TV
  Other Names: thoracic radiotherapy

SUMMARY:
This randomized phase III trial is studying carboplatin, paclitaxel, radiation therapy, and thalidomide to see how well they work compared to carboplatin, paclitaxel, and radiation therapy alone in treating patients with newly diagnosed stage III non-small cell lung cancer. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Thalidomide may stop the growth of non-small cell lung cancer by stopping blood flow to the tumor. It is not yet known if combination chemotherapy plus radiation therapy is more effective with or without thalidomide.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Compare the survival and time to progression of patients with stage IIIA or IIIB non-small cell lung cancer when treated with carboplatin, paclitaxel, and chemoradiotherapy with or without thalidomide.

II. Evaluate the toxicity of the thalidomide-containing regimen and compare response rates of the two groups.

III. Determine whether the inactivation of p16, Death-associated protein kinase (DAP-kinase), O6-methylguanine-DNA methyltransferase (MGMT) gene, or tissue-inhibitor of metalloproteinase 3 (TIMP-3) genes can be used to predict survival in these patients treated with this regimen.

IV. Determine whether the detection of a methylation biomarker in serum can be used to predict survival in these patients treated with this regimen.

OUTLINE: This is a randomized study. Patients are stratified according to disease histology (squamous vs nonsquamous), performance status (0 vs 1), disease stage (IIIA vs IIIB), and time of randomization (before addition of chemoradiotherapy vs after). Patients are randomized to one of two treatment arms.

ARM A: Patients receive paclitaxel intravenously (IV) over 3 hours immediately followed by carboplatin IV over 15-30 minutes on days 1 and 22. Treatment continues every 22 days in the absence of unacceptable toxicity or disease progression.

ARM B: Patients receive paclitaxel and carboplatin as in arm A. Patients also receive oral thalidomide and oral low-dose aspirin daily beginning on day 1 for up to 24 months in the absence of disease progression.

Beginning between days 43-50, patients in both arms with stable or responding disease receive chemoradiotherapy comprising paclitaxel IV over 1 hour and carboplatin IV over 15-30 minutes once weekly for 6 weeks and radiotherapy (RT) 5 days a week for 6 weeks. Arm B patients continue oral thalidomide.

Patients are followed every 2 months for 2 years and then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed newly diagnosed non-small cell bronchogenic carcinoma

  * Squamous cell
  * Adenocarcinoma
  * Large cell undifferentiated
  * Bronchoalveolar
  * Non-small cell carcinoma not otherwise stated
* Unresectable stage IIIA

  * Mediastinal lymph node enlargement of at least 1 cm but less than 2 cm on computed tomography (CT) scans must have mediastinotomy or thoracoscopy to rule out resectability

OR

* Stage IIIB disease without significant pleural effusion

  * Seen on CT scan only (not seen on chest x-ray) or does not reaccumulate after 1 thoracentesis and is cytologically negative
  * Metastases to contralateral, mediastinal, or supraclavicular nodes allowed
* Bidimensionally measurable or evaluable disease
* 18 and over
* ECOG performance status 0-1
* Adequate hematopoietic, hepatic, and renal function obtained <=4 weeks prior to registration:

  * Platelet count at least 100,000/mm^3
  * White Blood Cell (WBC) count at least 4,000/mm^3 OR absolute neutrophil count at least 2,000/mm^3
  * Bilirubin normal
  * Serum glutamic oxaloacetic transaminase (SGOT) no greater than 2.5 times upper limit of normal
  * Creatinine no greater than 1.5 mg/dL OR creatinine clearance at least 60 mL/min
* Fertile patients must use 2 methods of effective contraception for 4 weeks prior to, during, and for 4 weeks after study therapy
* Concurrent filgrastim (G-CSF) allowed for persistent neutropenia

Exclusion Criteria:

* Positive pregnancy test,pregnant or nursing
* Uncontrolled high blood pressure, unstable angina, congestive heart failure, or myocardial infarction within the prior year
* Serious cardiac arrhythmias requiring medication
* Prior radiotherapy to only area of measurable or active tumor
* Less than 5 years since prior chemotherapy
* Other active malignancies
* Serious uncontrolled active infection
* Evidence of greater than grade 1 neuropathy by history or physical examination
* History of seizure disorders
* Contraindication to daily low-dose (81 mg/day) aspirin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 589 (Actual)
Dates: Start 2000-01; Primary Completion 2009-12 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joan H. Schiller, MD, Study Chair — Simmons Cancer Center
Locations (236):
- United States (235):
  - Hembree Mercy Cancer Center at St. Edward Mercy Medical Center, Fort Smith, Arkansas
  - Memorial Medical Center Cancer Services, Modesto, California
  - Salinas Valley Memorial Hospital, Salinas, California
  - Stanford Comprehensive Cancer Center at Stanford University Medical Center, Stanford, California
  - Aurora Presbyterian Hospital, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Memorial Hospital, Colorado Springs, Colorado
  - Penrose Cancer Center at Penrose Hospital, Colorado Springs, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Presbyterian - St. Luke's Medical Center, Denver, Colorado
  - St. Joseph Hospital, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - CCOP - Colorado Cancer Research Program, Incorporated, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - St. Mary's Regional Cancer Center at St. Mary's Hospital and Medical Center, Grand Junction, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Hope Cancer Care Center at Longmont United Hospital, Longmont, Colorado
  - St. Mary-Corwin Regional Medical Center, Pueblo, Colorado
  - North Suburban Medical Center, Thornton, Colorado
  - Praxair Cancer Center at Danbury Hospital, Danbury, Connecticut
  - William W. Backus Hospital, Norwich, Connecticut
  - Halifax Medical Center - Daytona Beach, Daytona Beach, Florida
  - Baptist Cancer Institute - Jacksonville, Jacksonville, Florida
  - Veterans Affairs Medical Center - Augusta, Augusta, Georgia
  - MBCCOP - Medical College of Georgia Cancer Center, Augusta, Georgia
  - Veterans Affairs Medical Center - Atlanta (Decatur), Decatur, Georgia
  - Medical Center of Central Georgia, Macon, Georgia
  - Curtis & Elizabeth Anderson Cancer Institute at Memorial Health University Medical Center, Savannah, Georgia
  - Pearlman Comprehensive Cancer Center at South Georgia Medical Center, Valdosta, Georgia
  - Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois
  - Mercy Hospital and Medical Center, Chicago, Illinois
  - Swedish Covenant Hospital, Chicago, Illinois
  - Hinsdale Hematology Oncology Associates, Hinsdale, Illinois
  - Midwest Center for Hematology/Oncology, Joliet, Illinois
  - Trinity Medical Center - East, Moline, Illinois
  - Swedish-American Regional Cancer Center, Rockford, Illinois
  - Hematology/Oncology of the North Shore at Gross Point Medical Center, Skokie, Illinois
  - Elkhart General Hospital, Elkhart, Indiana
  - Howard Community Hospital at Howard Regional Health System, Kokomo, Indiana
  - Center for Cancer Therapy at LaPorte Hospital and Health Services, La Porte, Indiana
  - Reid Hospital & Health Care Services, Incorporated, Richmond, Indiana
  - CCOP - Northern Indiana CR Consortium, South Bend, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Saint Joseph Regional Medical Center, South Bend, Indiana
  - Hematology Oncology Associates of the Quad Cities, Bettendorf, Iowa
  - St. Luke's Hospital, Cedar Rapids, Iowa
  - Cedar Rapids Oncology Associates, Cedar Rapids, Iowa
  - Mercy Regional Cancer Center at Mercy Medical Center, Cedar Rapids, Iowa
  - Genesis Regional Cancer Center at Genesis Medical Center, Davenport, Iowa
  - Mercy Capitol Hospital, Des Moines, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Methodist Medical Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at John Stoddard Cancer Center, Des Moines, Iowa
  - Medical Oncology and Hematology Associates at Mercy Cancer Center, Des Moines, Iowa
  - Mercy Cancer Center at Mercy Medical Center - Des Moines, Des Moines, Iowa
  - John Stoddard Cancer Center at Iowa Lutheran Hospital, Des Moines, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Medical Oncology and Hematology Associates - West Des Moines, West Des Moines, Iowa
  - Merle M. Mahr Cancer Center at Regional Medical Center of Hopkins County, Madisonville, Kentucky
  - DeCesaris Cancer Institute at Anne Arundel Medical Center, Annapolis, Maryland
  - Tufts-NEMC Cancer Center, Boston, Massachusetts
  - Newton-Wellesley Hospital, Newton, Massachusetts
  - Baystate Regional Cancer Program at D'Amour Center for Cancer Care, Springfield, Massachusetts
  - Morton Hospital & Medical Center, Taunton, Massachusetts
  - Hickman Cancer Center at Bixby Medical Center, Adrian, Michigan
  - St. Joseph Mercy Cancer Center at St. Joseph Mercy Hospital, Ann Arbor, Michigan
  - CCOP - Michigan Cancer Research Consortium, Ann Arbor, Michigan
  - Oakwood Cancer Center at Oakwood Hospital and Medical Center, Dearborn, Michigan
  - Green Bay Oncology, Limited - Escanaba, Escanaba, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - Green Bay Oncology, Limited - Iron Mountain, Iron Mountain, Michigan
  - Foote Hospital, Jackson, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Borgess Medical Center, Kalamazooaa, Michigan
  - Haematology-Oncology Associates of Ohio and Michigan, PC, Lambertville, Michigan
  - Sparrow Regional Cancer Center, Lansing, Michigan
  - Mercy Memorial Hospital System, Monroe, Michigan
  - Seton Cancer Institute - Saginaw, Saginaw, Michigan
  - Lakeland Cancer Care Center at Lakeland Hospital - St. Joseph, Saint Joseph, Michigan
  - St. John Macomb Hospital, Warren, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - CCOP - Duluth, Duluth, Minnesota
  - Miller-Dwan Medical Center, Duluth, Minnesota
  - St. Mary's - Duluth Clinic Cancer Center, Duluth, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Fergus Falls, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Meeker County Memorial Hospital, Lichfield, Minnesota
  - HealthEast Cancer Care at St. John's Hospital, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center - Minneapolis, Minneapolis, Minnesota
  - Hubert H. Humphrey Cancer Center at North Memorial Medical Center, Robbinsdale, Minnesota
  - CentraCare Clinic - River Campus, Saint Cloud, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Health Services, Saint Louis Park, Minnesota
  - Regions Hospital Cancer Care Center, Saint Paul, Minnesota
  - St. Joseph's Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Cancer Center, Shakopee, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Woodwinds Health Campus, Woodbury, Minnesota
  - CCOP - Kansas City, Kansas City, Missouri
  - St. John's Regional Health Center, Springfield, Missouri
  - Hulston Cancer Center at Cox Medical Center South, Springfield, Missouri
  - Missouri Baptist Cancer Center, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - Deaconess Billings Clinic - Downtown, Billings, Montana
  - Big Sky Oncology, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Sletten Regional Cancer Institute at Benefis Healthcare, Great Falls, Montana
  - Great Falls, Montana
  - Cancer Resource Center - Lincoln, Lincoln, Nebraska
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Immanuel Medical Center, Omaha, Nebraska
  - Alegant Health Cancer Center at Bergan Mercy Medical Center, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - CCOP - Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Veterans Affairs Medical Center - East Orange, East Orange, New Jersey
  - Hunterdon Regional Cancer Center at Hunterdon Medical Center, Flemington, New Jersey
  - Cancer Institute of New Jersey at Hamilton, Hamilton, New Jersey
  - Fox Chase Virtua Health Cancer Program at Virtua Memorial Hospital Marlton, Marlton, New Jersey
  - Mountainside Hospital Cancer Center, Montclair, New Jersey
  - Carol G. Simon Cancer Center at Morristown Memorial Hospital, Morristown, New Jersey
  - Cancer Institute of New Jersey at UMDNJ - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Warren Hospital, Phillipsburg, New Jersey
  - Booker Cancer Center at Riverview Medical Center, Red Bank, New Jersey
  - Shore Memorial Hospital - Somers Point, Somers Point, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - Fox Chase Virtua Health Cancer Program at Virtua West Jersey, Voorhees Township, New Jersey
  - Veterans Affairs Medical Center - Buffalo, Buffalo, New York
  - Lipson Cancer and Blood Center at Rochester General Hospital, Rochester, New York
  - CCOP - Hematology-Oncology Associates of Central New York, Syracuse, New York
  - Albert Einstein Cancer Center at Albert Einstein College of Medicine, The Bronx, New York
  - Our Lady of Mercy Medical Center Comprehensive Cancer Center, The Bronx, New York
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Wilson Medical Center, Wilson, North Carolina
  - Bismarck Cancer Center, Bismarck, North Dakota
  - Cancer Care Center at Medcenter One Hospital, Bismarck, North Dakota
  - Mid Dakota Clinic, P. C., Bismarck, North Dakota
  - St. Alexius Medical Center, Bismarck, North Dakota
  - Akron City Hospital, Akron, Ohio
  - Aultman Hospital Cancer Center at Aultman Health Foundation, Canton, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - MetroHealth's Cancer Care Center at MetroHealth Medical Center, Cleveland, Ohio
  - Riverside Methodist Hospital Cancer Care, Columbus, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Grant Riverside Cancer Services, Columbus, Ohio
  - Mount Carmel Health - West Hospital, Columbus, Ohio
  - Doctors Hospital at Ohio Health, Columbus, Ohio
  - David L. Rike Cancer Center at Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Cancer Care Center, Dayton, Ohio
  - Veterans Affairs Medical Center - Dayton, Dayton, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Blanchard Valley Medical Associates, Findlay, Ohio
  - Fremont Memorial Hospital, Fremont, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - St. Rita's Medical Center, Lima, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - MedCentral - Mansfield Hospital, Mansfield, Ohio
  - Strecker Cancer Center at Marietta Memorial Hospital, Marietta, Ohio
  - St. Luke's Hospital, Maumee, Ohio
  - Northwest Ohio Oncology Center, Maumee, Ohio
  - Licking Memorial Cancer Care Program at Licking Memorial Hospital, Newark, Ohio
  - St. Charles Mercy Hospital, Oregon, Ohio
  - Firelands Regional Medical Center, Sandusky, Ohio
  - Mercy Medical Center, Springfield, Ohio
  - Community Hospital of Springfield and Clark County, Springfield, Ohio
  - Flower Hospital Cancer Center, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - Toledo Hospital, Toledo, Ohio
  - St. Vincent Mercy Medical Center, Toledo, Ohio
  - Medical University of Ohio Cancer Center, Toledo, Ohio
  - CCOP - Toledo Community Hospital, Toledo, Ohio
  - Toledo Clinic, Incorporated - Main Clinic, Toledo, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Morgan Cancer Center at Lehigh Valley Hospital - Cedar Crest, Allentown, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Oncology Hematology Associates of Northern Pennsylvania, PC at Hahne Regional Cancer Center, DuBois, Pennsylvania
  - Easton Regional Cancer Center at Easton Hospital, Easton, Pennsylvania
  - PinnacleHealth Regional Cancer Center at Polyclinic Hospital, Harrisburg, Pennsylvania
  - Penn State Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - Joan Karnell Cancer Center at Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Cancer Center at Phoenixville Hospital, Phoenixville, Pennsylvania
  - Allegheny Cancer Center at Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Hillman Cancer Center at University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - Pottstown Memorial Regional Cancer Center, Pottstown, Pennsylvania
  - Reading Hospital and Medical Center, Reading, Pennsylvania
  - Mercy Hospital Cancer Center - Scranton, Scranton, Pennsylvania
  - Hematology and Oncology Associates, Scranton, Pennsylvania
  - Grand View Hospital, Sellersville, Pennsylvania
  - Mount Nittany Medical Center, State College, Pennsylvania
  - Jennersville Regional Hospital, West Grove, Pennsylvania
  - Frank M. and Dorothea Henry Cancer Center at Geisinger Wyoming Valley Medical Center, Wilkes-Barre, Pennsylvania
  - CCOP - MainLine Health, Wynnewood, Pennsylvania
  - Lankenau Cancer Center at Lankenau Hospital, Wynnewood, Pennsylvania
  - Cancer Care Institute of Carolina at Aiken Regional Medical Centers, Aiken, South Carolina
  - CCOP - Greenville, Greenville, South Carolina
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Medical X-Ray Center, PC, Sioux Falls, South Dakota
  - Sioux Valley Hospital and University of South Dakota Medical Center, Sioux Falls, South Dakota
  - Christine LaGuardia Phillips Cancer Center at Wellmont Holston Valley Medical Center, Kingsport, Tennessee
  - MBCCOP - Meharry Medical College - Nashville, Nashville, Tennessee
  - CCOP - Scott and White Hospital, Temple, Texas
  - University of Virginia Cancer Center at UV Health System, Charlottesville, Virginia
  - Danville Regional Medical Center, Danville, Virginia
  - Southwest Virginia Regional Cancer Center, Norton, Virginia
  - Virginia Commonwealth University Massey Cancer Center, Richmond, Virginia
  - West Virginia University - Robert C. Byrd Health Sciences Center - Charleston Division, Charleston, West Virginia
  - Marshall University Medical Center, Huntington, West Virginia
  - Green Bay Oncology, Limited at St. Vincent Hospital, Green Bay, Wisconsin
  - Green Bay Oncology, Limited at St. Mary's Hospital, Green Bay, Wisconsin
  - St. Mary's Hospital Medical Center - Green Bay, Green Bay, Wisconsin
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Gundersen Lutheran Cancer Center at Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - Dean Medical Center - Madison, Madison, Wisconsin
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin
  - Bay Area Cancer Care Center at Bay Area Medical Center, Marinette, Wisconsin
  - Marshfield Clinic - Marshfield Center, Marshfield, Wisconsin
  - Green Bay Oncology, Limited - Oconto Falls, Oconto Falls, Wisconsin
  - All Saints Cancer Center at All Saints Healthcare, Racine, Wisconsin
  - Green Bay Oncology, Limited - Sturgeon Bay, Sturgeon Bay, Wisconsin
- Pretoria Academic Hospital, Pretoria, South Africa

REFERENCES:
- [Result] Belinsky SA, Grimes MJ, Casas E, Stidley CA, Franklin WA, Bocklage TJ, Johnson DH, Schiller JH. Predicting gene promoter methylation in non-small-cell lung cancer by evaluating sputum and serum. Br J Cancer. 2007 Apr 23;96(8):1278-83. doi: 10.1038/sj.bjc.6603721. Epub 2007 Apr 3. PMID 17406356
- [Result] Belinsky SA, Grimes M, Johnson D, et al.: Predicting gene promoter methylation in lung tumors through examination of sputum and serum. [Abstract] J Clin Oncol 24 (Suppl 18): A-7208, 416s, 2006.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was activated on January 27, 2000, and was terminated on October 26, 2006. 589 patients were enrolled to the study.
Groups:
- Arm A (Paclitaxel + Carboplatin + Radiation ): Active comparator. Induction dosing: Paclitaxel, 225 mg/m²; Carboplatin, AUC=6.0. Concurrent dosing: Paclitaxel, 45 mg/m2; Carboplatin: AUC=2.
- Arm B (Paclitaxel + Carboplatin + Radiation + Thalidomide): Experimental arm. Thalidomide: daily, patients begin with 200 mg thalidomide PO as a single dose at bedtime. The dose is then increased by 100 mg every week as tolerated up to a total dose of 1000 mg; low dose aspirin: 81mg PO daily.
  Paclitaxel, carboplatin and radiation same as active comparator.
Period: Overall Study
Arm/Group | Arm A (Paclitaxel + Carboplatin + Radiation ) | Arm B (Paclitaxel + Carboplatin + Radiation + Thalidomide)
Started | 295 | 294
Eligible | 275 | 271
Treated | 289 | 289
Treated and Having Toxicity Data | 289 | 288 (1 patient had missing record for toxicity)
Completed | 177 | 12
Not Completed | 118 | 282
Not completed — Lack of Efficacy | 43 | 113
Not completed — Adverse Event | 31 | 93
Not completed — Death | 5 | 5
Not completed — Withdrawal by Subject | 7 | 33
Not completed — Protocol Violation | 2 | 2
Not completed — other disease | 0 | 3
Not completed — error | 3 | 1
Not completed — missing data | 14 | 11
Not completed — Other | 13 | 21

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (Paclitaxel + Carboplatin + Radiation ) | Arm B (Paclitaxel + Carboplatin + Radiation + Thalidomide) | Total
Number analyzed (Participants) | 275 | 271 | 546
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.9 (9.0) | 62.2 (10.5) | 62.6 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 104 | 108 | 212
  Male | 171 | 163 | 334

OUTCOME MEASURES:

1. Secondary Outcome: Time to Disease Progression
Description: Time to disease progression is defined as the time from randomization to documented disease progression or to death without progression. Patients without documented progression or death reported were censored at the time of the last documented disease evaluation. Progression is defined, using the Response Evaluation Criteria In Solid Tumors (RECIST), as a measurable increase in the smallest dimension of any target or non-target lesion, or the appearance of new lesions, since baseline.
Time Frame: every other month until 24 months from study entry, every 3 months for year 3, every 4 months for the 4th year and every 6 months for the 5th year
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Arm A (Paclitaxel + Carboplatin + Radiation ): active comparator
- Arm B (Paclitaxel + Carboplatin + Radiation + Thalidomide): experimental arm
Arm/Group | Arm A (Paclitaxel + Carboplatin + Radiation ) | Arm B (Paclitaxel + Carboplatin + Radiation + Thalidomide)
Number analyzed (Participants) | 275 | 271
Months | 7.4 [6.6 to 8.6] | 7.8 [6.9 to 8.8]

2. Secondary Outcome: Response Rate at Best Response to Treatment
Description: Proportion of patients with complete or partial response using the Response Evaluation Criteria In Solid Tumors (RECIST) v1.0. Complete response is defined as the complete disappearance of all clinically detectable malignant disease for at least 4 weeks. Partial response is defined as greater than or equal to 50% decrease in tumor size for at least 4 weeks without increase in size of any area of known malignant disease of greater than 25%, or appearance of new areas of malignant disease.
Time Frame: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Arm A (Paclitaxel + Carboplatin + Radiation ) | Arm B (Paclitaxel + Carboplatin + Radiation + Thalidomide)
Number analyzed (Participants) | 275 | 271
Proportion of participants | 0.35 [0.29 to 0.41] | 0.38 [0.32 to 0.44]

3. Primary Outcome: Overall Survival Time
Description: Survival time is defined as time from study entry to death from any cause
Time Frame: every other month until 24 months from study entry, then every 3 months for year 3, every 4 months for year 4 and every 6 months for year 5
Population: intent to treat analysis in the 546 eligible patients
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A (Paclitaxel + Carboplatin + Radiation ) | Arm B (Paclitaxel + Carboplatin + Radiation + Thalidomide)
Number analyzed (Participants) | 275 | 271
Months | 15.3 [12.4 to 20.6] | 16.0 [14.5 to 18.5]
Statistical Analysis 1: Comparison: Arm A (Paclitaxel + Carboplatin + Radiation ) vs Arm B (Paclitaxel + Carboplatin + Radiation + Thalidomide); Test type: Superiority or Other; p = 0.99, Log Rank

ADVERSE EVENTS:
Time Frame: Toxicity assessment was conducted weekly during chemotherapy,every other month for 24 months during follow up, every 6 months once >24 months from study entry to 5 years.
Arm/Group | Arm A (Paclitaxel + Carboplatin + Radiation ) | Arm B (Paclitaxel + Carboplatin + Radiation + Thalidomide)
Serious Adverse Events (participants affected / at risk) | 222/289 | 249/288
Other Adverse Events (participants affected / at risk) | 283/289 | 284/288
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (Paclitaxel + Carboplatin + Radiation ) (N=289) | Arm B (Paclitaxel + Carboplatin + Radiation + Thalidomide) (N=288)
Allergic reaction (Immune system disorders) | 16 | 13
Inner ear/hearing imparied (Ear and labyrinth disorders) | 1 | 0
Hearing-other (Ear and labyrinth disorders) | 1 | 0
Anemia (Blood and lymphatic system disorders) | 8 | 4
Leukopenia (Investigations) | 69 | 81
Lymphopenia (Investigations) | 2 | 2
Neutropenia (Investigations) | 146 | 161
Thrombocytopenia (Investigations) | 10 | 6
Transfusion: platelets (Blood and lymphatic system disorders) | 1 | 0
Transfusion:pRBCs (Blood and lymphatic system disorders) | 15 | 6
Sinus bradycardia (Cardiac disorders) | 0 | 2
Sinus tachycardia (Cardiac disorders) | 1 | 1
Supraventricular arrhythmias (Cardiac disorders) | 2 | 6
Vasovagal episode (Nervous system disorders) | 1 | 0
Ventricular function (Cardiac disorders) | 2 | 1
Edema (General disorders) | 1 | 8
Hypertension (Vascular disorders) | 1 | 1
Hypotension (Vascular disorders) | 3 | 8
Pericardial effusion/pericarditis (Cardiac disorders) | 1 | 1
Peripheral arterial ischemia (Vascular disorders) | 0 | 1
Thrombosis/Embolism (Vascular disorders) | 6 | 30
Visceral arterial ischemia (Vascular disorders) | 0 | 1
Cardiac-other (Cardiac disorders) | 1 | 0
Fatigue (General disorders) | 16 | 42
Fever (General disorders) | 1 | 1
Weight gain (Investigations) | 0 | 1
Weight loss (Investigations) | 2 | 5
Elevated Partial Thromboplastin Time (PTT) (Investigations) | 1 | 0
Elevated Prothrombin Time (PT) (Investigations) | 0 | 1
Injection site reaction (General disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 4
Radiation dermatitis (Injury, poisoning and procedural complications) | 3 | 2
Rash/desquamation (Skin and subcutaneous tissue disorders) | 4 | 20
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 1
Wound -infectious (Injury, poisoning and procedural complications) | 0 | 1
Wound -non infectious (Injury, poisoning and procedural complications) | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 10 | 12
Constipation (Gastrointestinal disorders) | 4 | 26
Dehydration (Metabolism and nutrition disorders) | 10 | 6
Dyspepsia (Gastrointestinal disorders) | 3 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 2
Dysphagia-esophageal radiation (Injury, poisoning and procedural complications) | 4 | 3
Fistula-intestinal (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 2
Mucositis due to radiation (Injury, poisoning and procedural complications) | 1 | 0
Nausea (Gastrointestinal disorders) | 17 | 14
Stomatitis (Gastrointestinal disorders) | 8 | 7
Taste disturbance (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 14 | 7
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 5 | 8
GI-other (Gastrointestinal disorders) | 0 | 1
Melena/GI bleeding (Gastrointestinal disorders) | 0 | 1
Bilirubin increased (Investigations) | 0 | 1
AST increased (Investigations) | 1 | 0
ALT increased (Investigations) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 8 | 7
Infection w/ grade 3 or 4 neutropenia (Infections and infestations) | 9 | 15
Infection w/ unknown ANC (Infections and infestations) | 1 | 3
Infection w/o neutropenia (Infections and infestations) | 5 | 5
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 2
Hyperglycemia (Metabolism and nutrition disorders) | 8 | 4
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 1
Hypokalemia (Metabolism and nutrition disorders) | 3 | 11
Hyponatremia (Metabolism and nutrition disorders) | 14 | 15
Muscle weakness (Musculoskeletal and connective tissue disorders) | 2 | 3
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint,muscle, bone-other (Musculoskeletal and connective tissue disorders) | 0 | 1
Cerebrovascular Ischemia (Vascular disorders) | 0 | 2
Cognitive disturbance (Nervous system disorders) | 0 | 1
Confusion (Psychiatric disorders) | 0 | 2
Depressed level of consciousness (Nervous system disorders) | 1 | 15
Dizziness/lightheadedness (Psychiatric disorders) | 1 | 14
Hallucinations (Psychiatric disorders) | 0 | 2
Insomnia (Psychiatric disorders) | 1 | 0
Memory loss (Nervous system disorders) | 0 | 2
Depression (Psychiatric disorders) | 1 | 3
Neuropathy-motor (Nervous system disorders) | 5 | 9
Neuropathy-sensory (Nervous system disorders) | 16 | 33
Seizure (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 4 | 7
Tremor (Nervous system disorders) | 0 | 5
Vertigo (Ear and labyrinth disorders) | 1 | 2
Ocular-other (Eye disorders) | 0 | 1
Abonominal pain (Gastrointestinal disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 14
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 3
Chest pain (Cardiac disorders) | 2 | 2
Earache (Ear and labyrinth disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 7 | 14
Neuropathic pain (Nervous system disorders) | 2 | 0
Pain due to radiation (Injury, poisoning and procedural complications) | 2 | 2
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pain-other (General disorders) | 1 | 1
Apnea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 19 | 39
Hiccoughs (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 9
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 8 | 12
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Voice changes/dysarthria (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary - other (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Creatinine increased (Investigations) | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 0
Erectile impotence (Reproductive system and breast disorders) | 1 | 0
Irregular menses (Reproductive system and breast disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (Paclitaxel + Carboplatin + Radiation ) (N=289) | Arm B (Paclitaxel + Carboplatin + Radiation + Thalidomide) (N=288)
Leukopenia (Investigations) | 223 | 229
Anemia (Blood and lymphatic system disorders) | 238 | 238
Neutropenia (Investigations) | 187 | 220
Thrombocytopenia (Investigations) | 109 | 108
Edema (General disorders) | 24 | 83
Hypotension (Vascular disorders) | 18 | 31
Fatigue (General disorders) | 208 | 223
Fever (General disorders) | 20 | 15
Weight gain (Investigations) | 4 | 17
Weight loss (Investigations) | 79 | 64
Alopecia (Skin and subcutaneous tissue disorders) | 179 | 176
Dry skin (Skin and subcutaneous tissue disorders) | 7 | 25
Pruritus (Skin and subcutaneous tissue disorders) | 21 | 18
Radiation dermatitis (Injury, poisoning and procedural complications) | 58 | 55
Rash/desquamation (Skin and subcutaneous tissue disorders) | 49 | 89
Anorexia (Metabolism and nutrition disorders) | 110 | 97
Constipation (Gastrointestinal disorders) | 85 | 179
Dehydration (Metabolism and nutrition disorders) | 15 | 21
Dyspepsia (Gastrointestinal disorders) | 22 | 25
Dysphagia (Gastrointestinal disorders) | 25 | 30
Nausea (Gastrointestinal disorders) | 140 | 130
Stomatitis (Gastrointestinal disorders) | 58 | 68
Taste disturbance (Gastrointestinal disorders) | 47 | 54
Vomiting (Gastrointestinal disorders) | 68 | 50
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 62 | 40
Alkaline phosphatase increased (Investigations) | 62 | 56
AST increased (Investigations) | 34 | 19
Infection w/o neutropenia (Infections and infestations) | 27 | 28
Hyperkalemia (Metabolism and nutrition disorders) | 20 | 29
Hypokalemia (Metabolism and nutrition disorders) | 34 | 45
Hyponatremia (Metabolism and nutrition disorders) | 91 | 94
Depressed level of consciousness (Nervous system disorders) | 4 | 73
Dizziness/lightheadedness (Nervous system disorders) | 20 | 80
Insomnia (Psychiatric disorders) | 18 | 12
Anxiety/agitation (Psychiatric disorders) | 15 | 16
Depression (Psychiatric disorders) | 8 | 18
Neuropathy-motor (Nervous system disorders) | 34 | 60
Neuropathy-sensory (Nervous system disorders) | 161 | 206
Tremor (Nervous system disorders) | 3 | 31
Arthralgia (Musculoskeletal and connective tissue disorders) | 74 | 93
Headache (Nervous system disorders) | 28 | 35
Myalgia (Musculoskeletal and connective tissue disorders) | 110 | 117
Pain-other (General disorders) | 17 | 14
Cough (Respiratory, thoracic and mediastinal disorders) | 51 | 53
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 65 | 99
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 21 | 25
Creatinine increased (Investigations) | 27 | 32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less